CLINICAL TRIAL: NCT07063927
Title: The Impact of a Personalized Oral Health Instruction Form Health Indices in Institutionalized Older Adults: A Randomized, Controlled, Single-Blinded Clinical Trial.
Brief Title: Personalized Oral Hygiene Instruction Form
Acronym: POHIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Frauke Müller, Professeur, University of Geneva, Switzerland
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022-00086
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2023-06

CONDITIONS: Oral Hygiene, Oral Health; Plaque Score; Dental Plaque Index; Denture Hygiene; Tongue Coating Thickness
Keywords: oral hygiene; oral health; elderly; denture plaque score; dental plaque score; Tongue coating; medicalized homes; nursing homes

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The investigator conducting the oral examination was masked to the group allocation of the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): In the control group, both independent and dependent residents will receive a hygiene kit and verbal instructions on how to conduct care by the hygienist. Independent residents will perform their oral care themselves. Caregivers will provide oral care to dependent residents.
- intervention group (Active Comparator): In the intervention group, the participants will receive and oral hygiene kit along with the verbal instruction and in addition to that, they will also receive the written personalized oral instruction form by the second investigator, it will be displayed in the personal bathroom of the residents. For dependent residents, the personalized oral instruction form will be handed to the caregivers along with the personalized oral hygiene kit.
  Interventions: Procedure: personalized oral instruction form

INTERVENTIONS:
Procedure: personalized oral instruction form — The investigators will customize the POIF for participants. The POIF will be conceived to have a cover, and participants extraoral photos and intraoral photos will be covered when not conducting oral hygiene, the cover will ensure participants confidentiality. The personalized oral instruction form will be handed to the independent residents along with a hygiene kit comprising the necessary tools to conduct oral hygiene by the second investigator. For dependent residents, the personalized oral instruction form will be handed to the caregivers along with the personalized oral hygiene kit.
  Arms: intervention group

SUMMARY:
The objective of this study is to test a personalized oral hygiene instruction form (POHIF) elaborated after oral examination by a dentist and implemented by caregivers in nursing homes or similar medicalized homes.

DETAILED DESCRIPTION:
The study aims to test whether a newly developed tool can help caregivers improve the oral health indices of institutionalized residents.

Caregivers of the institution will be identified by the medicalized home and will be asked to answer a questionnaire pertaining to various aspects of oral health care. The questionnaire is divided into 5 themes, the first section will collect general information on the caregiver and will comprise 3 questions about age range, years of professional experience and current position. The investigators will not be able to identify the caregivers out of the 3 questions. The second theme will request information on the knowledge and clinical practices related to the oral care of dependent and independent in-residents. Caregivers will also rate the perceived importance of oral care in relation to general health on a Visual Analogue Scale (VAS) from 0 to 100. Other questions will inquire about tooth brushing, intraoral inspection, cleaning of prosthetic appliances and storage habits. The third theme consists of a closed check-list of instruments, asking if they were known to the caregivers and if they used it in their institutional setting. The fourth theme covers the caregivers' perception of oral care and potential barriers to its provision. The fifth and last theme related to the perceived barriers concerning institution logistics and resident-related factors. At the end of the fifth section, an open question will be added for a qualitative description of any additional barriers to oral care that were not covered by the previous questions.

The questionnaire will be filled in a focus group should the sanitary situation related to the pandemic permits; if necessary, the questionnaire can be administered online as well. The questionnaire will comprise 20 questions and one open ended question, and takes an average of 6-8 minutes to be completed. All caregivers in a unit will receive a theoretical oral health provision training, followed by a hands-on session. After the training, the caregivers will be asked to fill the same questionnaire and the answers/ scores will be compared before and after the training.

Resident living in an institution will be screened and included if fitting the inclusion and exclusion criteria. 46 participants will be recruited. After recruitment, all participants will receive an oral examination and an oral hygiene kit. The oral examination will record plaque index (PI) by O'Leary, denture cleanliness index (DCI) by Ambjornsen and tongue coating index (TCI) by Shimizu.

The participants will also be asked to fill a questionnaire about their own perception of their oral health related Quality of Life (General oral health assessment index, GOHAI). The oral examination will be conducted in the resident's room.

The investigators will then customize the POHIF for all participants. After the completion of all the examination in all recruited participants, participants then will be randomized into two groups. The randomization will be done in clusters according to the geographic location of the resident room so that bundles of rooms will be in one group and another bundle of rooms will be in another group. Investigators will ensure that the residents in the different units are not all dependent on care or independent and that they are representative of the institution population.

This bloc randomization will insure that participants that are in the same room belong to the same group. Randomization sequences will be obtained from www.randomizer.org. The sequences will be kept in sealed opaque envelopes.

The investigator that will conduct the first examination and elaborates the POIF will be blinded to the participant group allocation.

For participants in the intervention group, the personalized oral instruction form will be handed to the independent residents along with a hygiene kit comprising the necessary tools to conduct oral hygiene by the second investigator (N.M). For dependent residents, the personalized oral instruction form will be handed to the caregivers along with the personalized oral hygiene kit.

In the control group, independent and dependent residents will receive a hygiene kit, independent resident will continue to conduct their own oral care as usual, and for dependent residents, caregivers will provide the oral care as usual.

The duration of the study will be 3 weeks from the day of provision of the oral hygiene kit and the start of the intervention for every cluster of participants.

After 3 weeks, all included residents will get a second oral examination by the same investigator who conducted the first one.

Oral health indices will be again recorded.

ELIGIBILITY:
Inclusion Criteria:

* Living in an institution for more than 6 weeks
* Understand French
* Give written informed consent or consent can be obtained from their next of kin or legal representative if necessary

Exclusion Criteria:

* Non-cooperative participant
* Having an infectious disease (according to a medical report)
* Are undergoing currently dental treatment or need urgent treatment in next 3 weeks

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Plaque Index (PI) by O'Leary, Drake and Naylor | 3 weeks
  It is a simple, non-invasive plaque index utilizing visualization of deposits to assess a person's oral hygiene effectiveness. Plaque index is then calculated using the following formula: (the number of surfaces with plaque) / the total number of available tooth surfaces) x 100. PI percentages range from a minimum of 0% (i.e. no plaque on any tooth surface) to maximum of 100% (i.e. all remaining surfaces are covered by plaque).

SECONDARY OUTCOMES:
Denture cleanliness index modified (DCIM) by Ambjornsen | 3 weeks
  The present index was introduced to assess the location and amount of plaque in some areas of the fitting surfaces of complete maxillary dentures. Scores were recorded in five defined areas on the denture base. Four ranked scores were used:
  0: No visible plaque or plaque visible only by scraping on the denture base with a blunt instrument
  1: Moderate accumulation of visible plaque and abundance of plaque
Tongue coating index (TCI) by Shimizu | 3 weeks
  It is a visual method to assess the tongue-coating status based on observation of the coated thickness according 3 scores:
  Score 0: Tongue coating not visible Score 1: Tongue coating thin, papillae of tongue visible Score 2: Tongue coating very thick, papillae of tongue not visible

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Clinique universitaire de médecine dentaire, Geneva, Canton of Geneva
  - Maison de Vessy, Vessy, Canton of Geneva

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available upon reasonable request

REFERENCES:
- [Background] O'Leary TJ, Drake RB, Naylor JE. The plaque control record. J Periodontol. 1972 Jan;43(1):38. doi: 10.1902/jop.1972.43.1.38. No abstract available. PMID 4500182
- [Background] Shimizu T, Ueda T, Sakurai K. New method for evaluation of tongue-coating status. J Oral Rehabil. 2007 Jun;34(6):442-7. doi: 10.1111/j.1365-2842.2007.01733.x. PMID 17518979
- [Background] Ambjornsen E, Valderhaug J, Norheim PW, Floystrand F. Assessment of an additive index for plaque accumulation on complete maxillary dentures. Acta Odontol Scand. 1982;40(4):203-8. doi: 10.3109/00016358209019813. PMID 6958165
- [Derived] Chebib N, Rotzinger S, Maccarone-Ruetsche N, Sioufi R, Mojon P, Muller F. The impact of a personalized oral health instruction form on oral health indices in institutionalized older adults: a randomized, controlled, single-blinded clinical trial. BMC Oral Health. 2025 Nov 10;25(1):1769. doi: 10.1186/s12903-025-07102-y. PMID 41214684